CLINICAL TRIAL: NCT06764511
Title: Valutazione Della Risposta Alla Terapia Con Eritropoietina Alfa Biosimilare Nei Pazienti Anemici Affetti da Sindrome Mielodisplastica
Brief Title: Evaluation of Response to Biosimilar Erythropoietin Alfa Therapy in Anemic Patients With Myelodysplastic Syndrome
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EPO BIOSIM
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to describe the response to treatment with biosimilar EPO alpha in MDS patients who had already been treated with "originator" EPO alpha and were responsive, and in patients who started treatment with biosimilar EPO alpha

DETAILED DESCRIPTION:
To date, therapy with erythropoiesis-stimulating agents (ESAs) has been shown to be effective in the treatment of symptomatic anemia in patients with Myelodysplastic Syndrome ( MDS) at low to intermediate risk, with the percentage of responsive patients ranging from 15 to 63%, depending on the characteristics of the patients treated, and averaging 45%.

Significant improvement in survival and quality of life was observed in treatment-responsive patients compared with non-responsive patients.

Recently, biosimilar ESAs have been introduced into clinical practice, and in patients with renal failure anemia and anemia associated with antineoplastic chemotherapy, their efficacy and safety have been demonstrated.

However, data on the efficacy and safety of biosimilar ESAs in patients with MDS are scarce to date, and efficacy and safety data for the purpose of their approval have been mainly extrapolated from studies conducted in patients with anemia from renal failure and anemia from antineoplastic chemotherapy. In these conditions bone marrow erythropoiesis is reduced but not qualitatively impaired as in MDS.

These considerations may justify a retrospective study examining the efficacy and safety of biosimilar EPO alpha in a real-life setting in anemic MDS patients.

ELIGIBILITY:
Inclusion Criteria:

MDS patients with symptomatic anemia (pre-treatment hemoglobin < 10g/dL) who started treatment with biosimilar EPO alpha, diagnosed according to the WHO 2016 classification, and characterized by very low, low, or intermediate IPSS-R risk and a pre-treatment serum EPO level < 500 U/L, who started treatment with biosimilar EPO alpha at the U. O. of Hematology of IRCCS AOUBO during the period from 01/06/2018 to 31/12/2021.

* Age ≥ 18 years at the time of enrollment
* Acquisition of informed consent to study participation and data processing

Exclusion Criteria:

* - Presence of other possible contributory causes of anemia (e.g., anemia from chronic inflammatory disease, hemolysis, hemorrhage)
* Poor compliance with treatment
* Very impaired general clinical condition (ECOG performance status > 3)
* Concomitant treatment with antineoplastic cytotoxic drugs

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with MDS who started treatment with biosimilar EPO alpha at the "Seràgnoli" Institute, U.O. of Hematology of IRCCS AOU of Bologna during the period from 01 Jun 2018 to 31 Dec 2021 will be enrolled in the study.
  Specifically, the population will consist of
  * patients who initiated treatment after having already been treated with "originator" EPO alfa and responsive to treatment at the time of initiation of biosimilar EPO alfa, and
  * patients who started treatment without previous treatment with biosimilar EPO alfa
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Response and maintenance of ORR | 6 months from the start of the study
  response to treatment (ORR) (assessed according to the response criteria established by the International Working Group (23) in patients who initiated treatment with biosimilar EPO alfa
  - maintenance of ORR (assessed according to the response criteria established by the International Working Group (23) from the date of biosimilar drug initiation), in patients previously on treatment and responsive to "originator" EPO alfa who were subsequently treated with biosimilar EPO alfa

SECONDARY OUTCOMES:
A measure of the frequency of major clinical outcomes in two groups of patients who had different modes of treatment administration with biosimilar EPO alpha | 6 months from the start of the study
  1) DOR to EPO alpha: to biosimilar drug only in patients who started treatment with biosimilar EPO alpha; to "originator" drug + biosimilar in patients already on treatment and responsive to "originator" EPO alpha who were subsequently treated with biosimilar EPO alpha ; 2) incidence of adverse events in year/person (in both patient groups) according to NCI-CTCAE v.5.0 ; 3) number of patients who discontinued treatment with the biosimilar drug due to intolerance, loss of response, disease progression (DP), evolution into AML, or death (both groups) ; 4) number of patients who resumed the originator drug due to intolerance or failure to respond to the biosimilar drug ; 5) ORR and incidence of adverse events of patients who resumed treatment with "originator" EPO alfa after discontinuation of the biosimilar drug ; 6) incidence of evolution into AML in year/person (both groups) ; 7) OS and causes of death (both groups)

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Paolini, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliera -Universitaria di Bologna, Bologna, Italy